CLINICAL TRIAL: NCT05520177
Title: A Randomized, Double Masked, Multicenter, Phase III Study Assessing the Efficacy and Safety of 601 Versus Ranibizumab in Patients With Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Brief Title: A Phase III Study for 601 Versus Ranibizumab in Patients With Vision Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-601-BRVO-III-01
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2023-01

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: Retinal Vein Occlusion; Macular Edema; Vascular Endothelial Growth Factor
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 601 1.25mg (Experimental): loading phase (6 months): 601 1.25mg/eye/time, Intravitreal injection, administered once every 4 weeks for 6 consecutive doses
  Interventions: Drug: 601 1.25mg
- ranibizumab 0.5mg (Active Comparator): loading phase (6 months): ranibizumab 0.5mg/eye/time, Intravitreal injection, administered once every 4 weeks for 6 consecutive doses
  Interventions: Drug: ranibizumab 0.5mg

INTERVENTIONS:
Drug: 601 1.25mg — loading phase (6 months): 601 1.25mg/eye/time, Intravitreal injection, administered once every 4 weeks for 6 consecutive doses
  Other Names: 601
  Arms: 601 1.25mg
Drug: ranibizumab 0.5mg — loading phase (6 months): ranibizumab 0.5mg/eye/time, Intravitreal injection, administered once every 4 weeks for 6 consecutive doses
  Other Names: Lucentis
  Arms: ranibizumab 0.5mg

SUMMARY:
To compare the efficacy and safety of recombinant humanized anti-VEGF monoclonal antibody (601) with Ranibizumab in patients with macular edema secondary to BRVO

DETAILED DESCRIPTION:
After a up to 14-day screening period, patients will be randomized allocated in 2 groups at 1:1 ratio and followed up for 52 weeks. Followed-up visits will be scheduled at a 4-week interval. After 6 initial monthly injections of 601 or ranibizumab (loading phase), subjects will enter an individualized flexible treatment (IFT) phase (week 24 to week 48). During the IFT phase, subjects will receive either the injections or not based on the assessment of disease stability at each visit. Efficacy and safety outcomes will be evaluated up to a period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form and willing to be followed up at the time specified in the trial
* Male or Female, at least 18 years of age
* The study eye must meet the following criteria：Diagnosed with macular edema secondary to Branch retinal vein occlusion (BRVO) or Hemi-retinal vein occlusion (HRVO) within 12 months; BCVA score ≤ 73 and ≥19 letters using ETDRS visual acuity testing charts (approximate Snellen equivalent of 20/40 to 20/400); CRT ≥ 250μm; No optometric media opacity and pupil abnormal
* BCVA score ≥ 34 ETDRS letters (approximate Snellen equivalent of 20/200) in the fellow eye, with no active RVO disease.

Exclusion Criteria:

* For Study Eye: Concomitant conditions or ocular disorders in the study eye at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the 52-week study period
* For Study Eye: iris, chamber angle neovascularization or retinal, optic disc neovascularization
* For Study Eye: Previous use of intraocular or periocular steroids within 3 months prior to baseline, or dexamethasone intravitreal implant within 6 months prior to baseline
* For Study Eye: Macular laser photocoagulation (focal/grid)，panretinal laser photocoagulation，vitrectomy，trabeculectomy or keratoplasty in the study eye at any time prior to baseline. YAG laser treatment or any other intraocular surgeries (e.g. cataract surgery) in the study eye within 3 months prior to the baseline
* For Study Eye: During the screening period, the BCVA is >10 letters improved
* For Study Eye: Aphakia (except IOL) or posterior capsular defect (except YAG posterior capsulotomy after intraocular lens implantation surgery)
* For Any Eye: Active ocular infections (e.g. blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in any eye
* For Any Eye: Uncontrolled glaucoma (defined as intraocular pressure after antiglaucoma therapy ≥ 25mmHg) in any eye, or the cup/disk ratio >0.8 in the study eye
* For Any Eye: History of intravitreal use of anti-VEGF drugs (e.g. ranibizumab，bevacizumab，aflibercept, conbercept, etc.) in any eye within 3 months prior to baseline
* History of allergy to fluorescein sodium and allergies to protein products for treatment or diagnosis
* History of stroke (cerebrovascular accident), myocardial infarction, active disseminated intravascular coagulation or pronounced bleeding tendency in the past 6 months prior to baseline
* Systemic immune diseases (e.g. ankylosing spondylitis, systemic lupus erythematosus, Behcet's disease, rheumatoid arthritis, scleroderma etc.)
* Any uncontrolled clinical conditions (e.g. AIDS, active hepatitis, serious mental, neurological, cardiovascular, respiratory and other systemic diseases or malignant tumors, etc.). Malignant tumors with no metastasis or recurrence within 5 years or cancers in situ cancers are not excluded.
* Uncontrolled blood pressure (defined as systolic blood pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg after antihypertensive medication
* History of surgery (except for healed minimally invasive surgery) and/or currently have unhealed wounds, moderate to severe ulcers, fractures, etc. within 1 month prior to baseline
* History of system use of anti-VEGF drugs (e.g. bevacizumab) within 3 months prior to baseline
* Liver dysfunction (ALT or AST is 2 times higher than the upper limit of normal value in the local laboratory). Renal function impairment (Cr is 1.5 times higher than the upper limit of normal values in the local laboratory)
* Abnormal coagulation function (prothrombin time ≥ the upper limit of normal value for 3 seconds) and activated partial thromboplastin time ≥ the upper limit of normal value for 10 seconds).
* Non-use of effective contraception during childbearing age (except for women with spontaneous admonishment of more than 12 months)
* Women in pregnancy and lactation
* Participation in clinical trials of any drug (except vitamins and minerals) or medical devices in the past 1 month or 5 half-lifes if the drug has a long half-life >1 month prior to baseline.
* Any conditions that researchers think it needs to be ruled out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
best-corrected visual acuity (BCVA) | From Baseline to Week 24
  Assessed with Early treatment diabetic retinopathy study (ETDRS) visual acuity testing charts.

SECONDARY OUTCOMES:
best-corrected visual acuity (BCVA) | up to 52 weeks
  Assessed with Early treatment diabetic retinopathy study (ETDRS) visual acuity testing charts.
central retinal thickness (CRT) | up to 52 weeks
  SD-OCT (spectral domain optical coherence tomography) was used to assess the average retinal thickness of the central 1 mm diameter subfield around the foveal center.
Number of injections | up to 52 weeks
  Number of administered injections for 601 or ranibizumab
Adverse Events (AEs) | up to 52 weeks
  All adverse events related to 601 or ranibizumab observed through various tests (including blood routine, pregnancy test, electrocardiogram, etc.)
Steady-state Blood concentrations of 601 or ranibizumab | up to 52 weeks
  Detect the steady-state blood concentrations of 601 or ranibizumab through the subject's blood sample
Blood concentrations of Vascular Endothelial Growth Factor (VEGF) | up to 52 weeks
  Detect the blood concentrations of VEGF through the subject's blood sample
anti-drug antibody (ADA) of 601 | up to 52 weeks
  Detect the presence of anti-drug antibody (ADA) of 601 through the subject's blood sample. ADA-positive subjects will also undergo further Neutralization antibody (Nab) testing.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, MD, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (10):
- China (10):
  - BeiJing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of JiNan University, Guangzhou, Guangdong
  - HeNan Provincial Eye Hospital, Zhengzhou, Henan
  - The Second XiangYa Hospital of Central South University, Changsha, Hunan
  - JiangSu Province Hospital, Nanjing, Jiangsu
  - ShangHai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - TianJin Eye Hospital, Tianjin, Tianjin Municipality
  - TianJin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - ZheJiang Province People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No